CLINICAL TRIAL: NCT01642108
Title: The Effect of Sitagliptin, a Dipeptidyl Peptidase-4 Inhibitor, on Glycemic Control and Inappropriate Glucagon Secretion in Non-obese Japanese Patients With Type 2 Diabetes.
Brief Title: Treatment With Sitagliptin in Non-obese Japanese Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Niigata Medical Center (Other)
Collaborators: Nagaoka Red Cross Hospital (Other)
Responsible Party: Principal Investigator, Nobumasa Ohara, Principal Investigator, Niigata Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-Ohara
Record Dates: First submitted 2012-06-07; First posted 2012-07-17 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sitagliptin (Other)
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — 50 mg once per day
  Other Names: Other name is known

SUMMARY:
Type 2 diabetes mellitus (T2DM) results from early phase insulin secretory defect and insulin resistance. Studies have shown that most of the populations in which insulin resistance is considered to be the primary pathogenetic cause of diabetes, have a higher degree of obesity than those of primary insulin defect. Meanwhile, defective early insulin secretion plays a predominant role in the non-obese subtype of T2DM which includes majority of Japanese patients.

Sitagliptin is a dipeptidyl peptidase-4 (DPP-IV) inhibitor as indicated for the treatment of T2DM. Sitagliptin increases plasma concentrations of active glucagon-like peptide-1 (GLP-1) and active glucose-dependent insulinotropic peptide (GIP) two- to three-fold in patients with T2DM. The effect of sitagliptin on GLP-1 results in lower fasting and postprandial glucose concentrations through increases in glucose dependent insulin release and suppression of inappropriate glucagon secretion. Namely, several mechanistic studies using standardized meal showed that sitagliptin improved glucose control with decreased glucagon levels and increased insulin concentration in obese or overweight T2DM patients with BMI > 25 kg/m2. However, how sitagliptin affects islet function, including glucagon secretion in non-obese patients with low insulin secretion are not known. Therefore, the investigators will examine the effect of sitagliptin on glycemic control and the mechanism involved using a standardized test meal in non-obese Japanese patients with T2DM whose BMI levels are < 25 kg/m2.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients
* non-obese patients

Exclusion Criteria:

* patients treated with insulin therapy
* patients aged less than 20 years and more than 90 years

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-05 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
HbA1c | One month

SECONDARY OUTCOMES:
Glucagon secretion | One month

CONTACTS AND LOCATIONS:
Locations (1):
- Nobumasa Ohara, Niigata, Niigata, Japan